CLINICAL TRIAL: NCT06338839
Title: Multicenter Observational Retrospective-prospective Study of Prevalence and Clinical Characteristics of Transthyretin Amyloidosis Cardiomyopathy in Russian Patients With Heart Failure With Preserved Ejection Fraction in Real Clinical Practice
Brief Title: Transthyretin Amyloidosis Cardiomyopathy in Patients With HFpEF in Russia
Acronym: TETRAMER
Status: Terminated | Type: Observational
Why Stopped: The study was suspended after interim analysis to confirm reasonability of further investigation of the population
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8450R00006
Record Dates: First submitted 2024-03-04; First posted 2024-04-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Transthyretin Amyloidosis Cardiomyopathy, Heart Failure With Preserved Ejection Fraction
Keywords: Transthyretin amyloidosis cardiomyopathy, heart failure with preserved ejection fraction, ATTR, CM, HFpEF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter observational retrospective-prospective study of prevalence and clinical characteristics of transthyretin amyloidosis (ATTR) cardiomyopathy (CM) in Russian patients with heart failure with preserved ejection fraction (HFpEF) in real clinical practice.

The retrospective phase will entail secondary data collection from electronic or paper medical records of patients who are participating/participated in the PRIORITY-CHF study and have HFpEF. Those patients who have a high suspicion of having ATTR-CM and provided informed consent will be invited to participate in the prospective phase. The prospective phase will consist of three visits, during which a routine comprehensive cardiologic evaluation in order to confirm or exclude ATTR-CM diagnosis will be performed. In patients with confirmed ATTR-CM the material for genetic testing will be collected in order to specify the type of ATTR-amyloidosis

DETAILED DESCRIPTION:
This is a multicenter observational study consisting of retrospective and prospective phases.

Heart failure (HF) - is a clinical syndrome characterised by the presence of typical symptoms (e.g. breathlessness, fatigue and ankle swelling) and signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral oedema) caused by a structural and/or functional cardiac abnormality, resulting in a reduced cardiac output and/or elevated intracardiac pressures at rest or during stress.

Cardiac amyloidosis is an underestimated cause of HF and cardiac arrhythmias. Among all most commonly types of cardiac amyloidosis (wild-type or familial TTR and light-chain), the wild-type (Wt) TTR-related amyloidosis (ATTR) is an increasingly recognized cause of HFpEF, and amyloidosis should be considered in the differential diagnosis of this heart failure group of patients.

ATTR-CM is an inexorably progressive and eventually fatal, associated with poor quality of life. Diagnosis is often delayed for many years after symptoms develop. However, recognition of ATTR epidemiology is evolving due to the increased use of cardiac scintigraphy as a noninvasive diagnostic tool. Early identification and intervention are crucial to improve patient outcomes because newly available treatments have been shown to have maximum therapeutic benefit when started in the early stages of the disease. In recent years, contemporary cardiac imaging techniques, including MRI and bone scintigraphy, have altered the diagnostic algorithm for ATTR-CM, which has resulted in increased detection.

Thus country-specific epidemiologic data collection and identification of ATTR-CM is crucial to improve outcomes and quality of life. However, no observational studies on the epidemiology of ATTR-CM in Russian patients with HFpEF have been performed.

Therefore, there is a need to conduct a large-scale observational study to determine the prevalence of ATTR-CM in Russia, obtain information on patients' clinical characteristics, and determine their medical needs. Meanwhile information about epidemiological, ECG, EchoCG, other characteristics and prevalence is crucially important to improve diagnostics of these patients.

In addition, recently molecular genetic testing became available, which is essential to diagnose hereditary ATTR. Earlier recognition of the ATTR type, in turn, may lead to timely treatment initiation and change in the prognostic outlook of ATTR-CM patients.

ELIGIBILITY:
Inclusion Criteria:

for the retrospective phase are:

* Patients participating/participated in the PRIORITY-CHF study (may be alive or deceased at the time of inclusion to this study).
* Established diagnosis of HFpEF (presence of typical signs and symptoms of HF (see Appendix A) and LVEF ≥50%) at any time during participation in the PRIORITY-CHF study.

The following criteria apply for inclusion of patients into the prospective part of the study:

* Provided written informed consent for the prospective phase of the study.
* Presence of left ventricular wall thickness >12 mm.
* Presence of at least three of "red flags" or additional signs for having high-risk of ATTR-CM (evaluation based on medical history of HF and concomitant diseases, family history, results of previous ECG, Echo-CG/cardiac MRI, laboratory data):

  * >65 age (during participation in the PRIORITY-CHF study)
  * Conduction system disease (atrioventricular block, left bundle branch block, long QRS complex, sick sinus syndrome)/pacemaker
  * Atrial fibrillation
  * Pseudoinfarct pattern on the ECG (when hemodynamically significant stenosis is absent);
  * Disproportion of QRS voltage to the degree of increased LV wall thickness on imaging methods
  * Grade 2 or worse diastolic dysfunction
  * Decreased longitudinal strain with apical sparing
  * Diffuse subendocardial or transmural late gadolinium enhancement on cardiac MRI with increased extracellular volume fraction
  * Persistent low-level troponin elevation
  * Elevated NT-proBNP level
  * Right ventricular (RV) wall thickness more than 6 mm
  * Pericardial effusion in patients with LV-hypertrophy
  * Restrictive pattern in patients with LV-hypertrophy
  * Atrial enlargement with the normal ventricular volumes
  * Bilateral carpal tunnel syndrome
  * Lumbar/cervical spinal stenosis
  * Spontaneous biceps tendon rupture
  * Hip or knee replacement
  * Peripheral neuropathy
  * Family history of neuropathy
  * Intolerance/poor tolerance to vasodilating antihypertensive medications
  * Orthostatic hypotension
  * Gastroparesis
  * Urinary incontinence (neurogenic bladder), recurrent urinary infections,
  * Erectile dysfunction
  * Other autonomic dysfunction, such as gastrointestinal motility disorders (constipation, early satiety, chronic diarrhea, nausea/vomiting), syncope, anhidrosis)

Exclusion Criteria:

Exclusion criteria for the retrospective phase are:

* Any severe condition that, in opinion of the physician, will limit patient's life span to 12 months or less from the inclusion to this study.
* Current participation in any interventional trial (i.e. at the time of inclusion to this study).

The following criteria apply for exclusion of patients from the prospective part of the study:

* Patients with previously established (and documented) ATTR-CM.
* Patients with previous positive hematological test result on evaluating AL-amyloidosis in the anamnesis (monoclonal protein is identified by SIFE/UIF) and the serum FLC ratio (kappa/lambda) is in outside of the normal range).

If the hematological test on evaluating AL amyloidosis is negative, or there is no such test performed in the patient's medical history, the patient may be enrolled to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned study population consists of approximately 6000 patients with HFpEF who are participating/participated in the PRIORITY-CHF study and will be enrolled to this study across 140 clinical centers in different regions of Russia, in order to provide a representative study sample. Those patients who have a high suspicion of having ATTR-CM and provided informed consent will be invited to participate in the prospective phase. The patients will be included to the current study consecutively, from the earliest date of start of participation in the PRIORITY-CHF study.
Sampling Method: Non-Probability Sample
Enrollment: 1770 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of ATTR-CM in patients with HFpEF in routine clinical practice in the Russian Federation | Up to 12 months
  In order to achieve primary objective, the proportion of patients with confirmed diagnosis of ATTR-CM (at the end-of-study visit, according to the results of comprehensive cardiologic examination) among patients with HFpEF who were enrolled to retrospective phase and prospective phase of this study will be calculated.

SECONDARY OUTCOMES:
demographic and clinical characteristics, and test results | Up to 12 months
  In order to achieve the secondary objectives, the following demographic and clinical characteristics, and test results (with additional available data as needed) will be assessed in patients who were enrolled to the prospective phase of this study: Mean age (years) at the diagnosis of HFpEF during participation in the PRIORITY-CHF study; Mean age at the diagnosis of ATTR-CM confirmed in this study (assessed in patients with confirmed ATTR-CM); Mean and median time from the diagnosis of HFpEF to the confirmed diagnosis of ATTR-CM (assessed in patients with confirmed ATTR-CM); Distribution of patients by age group sex, race, ethnicity and geographic regions; Mean body mass index (BMI) and proportion of patients with different BMI dimensions; Proportion of patients with a history of unexplained weight loss (≥5 kg) at any point; Mean blood pressure (BP) and heart rate; Proportion of patients with presence of negative lifestyle factors (smoking and alcohol abuse); etc.

CONTACTS AND LOCATIONS:
Locations (21):
- Russia (21):
  - Research Site, Akhtubinsk
  - Research Site, Astrakhan
  - Research Site, Barnaul
  - Research Site, Beslan
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Khabarovsk
  - Research Site, Kirov
  - Research Site, Krasnodar
  - Research Site, Nizhny Novgorod
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Smolensk
  - Research Site, Ufa
  - Research Site, Vladimir
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8450R00006&attachmentIdentifier=2039ab7b-94f2-4d9d-8dbb-b30f092ae6a7&fileName=D8450R00006_Study_interim_report_Synopsis_Redacted.pdf&versionIdentifier=